CLINICAL TRIAL: NCT04359303
Title: Randomized Clinical Trial to Evaluate Efficacy and Safety of Systemic Indirect Endovenous Ozone Therapy (SIEVOT) as Adjuvant Treatment in COVID19 Non-intubated Patients
Brief Title: Indirect Endovenous Systemic Ozone for New Coronavirus Disease (COVID19) in Non-intubated Patients
Acronym: OzonoCOVID19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Javier Hidalgo Tallón (Other)
Collaborators: Sociedad Española de Ozonoterapia (Other)
Responsible Party: Sponsor-Investigator, Javier Hidalgo Tallón, Lecturer, Universidad Católica San Antonio de Murcia
Organization: Universidad Católica San Antonio de Murcia (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P.Inv. Ozono-COVID19 Ver.1.2
Record Dates: First submitted 2020-04-09; First posted 2020-04-24 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: COVID
Keywords: ozone therapy; COVID19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Control group with WHO recommended treatment. Treatment group with WHO recommended treatment + systemic ozone therapy.
Who Masked: Participant, Investigator
Masking Description: With a randomization table, nurses will treat the patients in treatment groups. Each patient will be in individual rooms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (No Intervention): Base WHO recommended treatment.
- TREATMENT (Experimental): Base WHO recommended treatment + Systemic indirect endovenous ozone therapy
  Interventions: Other: Systemic indirect endovenous ozone therapy

INTERVENTIONS:
Other: Systemic indirect endovenous ozone therapy — 200 mL at 40 mcg/mL of medical ozone / oxygen in 200 mL of patients blood mixed in an homologated device for the procedure.
  Arms: TREATMENT

SUMMARY:
Systemic medical ozone has proved to help in several viral diseases, chronic obstructive pulmonary disease and chronic inflammation process. The investigators are sure that its application to COVID-19 patients, as an adjuvant therapy, will improve the health status of these individuals.

DETAILED DESCRIPTION:
Due to the extreme world situation caused by COVID19 pandemic, the investigators consider unethical not to try any treatment option with a justified rationale.

The investigators have explained that medical ozone therapy has a clear scientific basement thanks to all preclinical and clinical investigation already published. It can be classified as chemical stressor that produces a modulation in the redox balance and immunity. Moreover, it is easy and safe to administer with insignificant side effects.

The efficacy in viral diseases has been proved in publications together the modulation of interleukin 6 and other proinflammatory cytokines that could potentially help in COVID19 patients. The improve of exchange of gases and microcirculation will surely contribute to enhance this patients' health status.

As explained above, the investigators propose to carry out a randomized control trial to evaluate the safety and efficacy of systemic ozone (indirect endovenous) in these patients.

ELIGIBILITY:
Inclusion Criteria:

* COVID19 virus detected in oro/nasopharynx
* mild ill according WHO numeric scale
* mild ill according Berlin criteria
* non intubated patients
* signed informed consent

Exclusion Criteria:

* patients treated with systemic ozone in the last 6 months
* patients treated before with systemic ozone and referring any side effect
* glucose-6-phosphate-dehydrogenase deficit
* other severe concomitant disease apart from COVID19
* psychiatric disease specified in axis I of l Diagnostic and Statistical Manual of Mental Disorders, 5 edition, but major depression
* patients not capable of understanding the study methods and targets
* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
COVID19 clinical scale | through study completion, an average of 3 weeks
  World Health Organization (WHO) recommended COVID19 clinical scale

SECONDARY OUTCOMES:
Number of died patients | through study completion, an average of 3 weeks
  Dead patients during the trial
Oro/nasopharynx virus | through study completion, an average of 3 weeks
  Oro/nasopharynx virus
Thorax imaging (0=none; 1=unilateral; 2=bilateral; 3=ground-glass opacification; 4=consolidation) | through study completion, an average of 3 weeks
  Thorax imaging according scale. Higher punctuation is worse.
Days in hospital | through study completion, an average of 3 weeks
  Days in hospital
Venous gas blood analysis | through study completion, an average of 3 weeks
  Venous gas blood analysis

CONTACTS AND LOCATIONS:
Locations (1):
- SEOT, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
According to hospitals' statements and data protection agreements

REFERENCES:
- [Background] Bocci V. Ozone: A new medical drug. Netherlands: Springer; 2011.
- [Background] Baeza J, Cabo JR, Gómez M, et al. WFOTs Review on Evidence Based Ozone Therapy. World Federation of Ozone Therapy. Brescia: WFOT; 2015.
- [Background] Bocci V, Valacchi G. Nrf2 activation as target to implement therapeutic treatments. Front Chem. 2015 Feb 2;3:4. doi: 10.3389/fchem.2015.00004. eCollection 2015. PMID 25699252
- [Background] Pecorelli A, Bocci V, Acquaviva A, Belmonte G, Gardi C, Virgili F, Ciccoli L, Valacchi G. NRF2 activation is involved in ozonated human serum upregulation of HO-1 in endothelial cells. Toxicol Appl Pharmacol. 2013 Feb 15;267(1):30-40. doi: 10.1016/j.taap.2012.12.001. Epub 2012 Dec 16. PMID 23253326
- [Background] Re L, Martinez-Sanchez G, Bordicchia M, Malcangi G, Pocognoli A, Morales-Segura MA, Rothchild J, Rojas A. Is ozone pre-conditioning effect linked to Nrf2/EpRE activation pathway in vivo? A preliminary result. Eur J Pharmacol. 2014 Nov 5;742:158-62. doi: 10.1016/j.ejphar.2014.08.029. Epub 2014 Sep 16. PMID 25218903
- [Background] Hernandez Rosales FA, Calunga Fernandez JL, Turrent Figueras J, Menendez Cepero S, Montenegro Perdomo A. Ozone therapy effects on biomarkers and lung function in asthma. Arch Med Res. 2005 Sep-Oct;36(5):549-54. doi: 10.1016/j.arcmed.2005.04.021. PMID 16099337
- [Background] Calunga JL, Paz Y, Menendez S, Martinez A, Hernandez A. [Rectal ozone therapy for patients with pulmonary emphysema]. Rev Med Chil. 2011 Apr;139(4):439-47. Epub 2011 Aug 25. Spanish. PMID 21879181
- [Background] Borrelli E, Bocci V. Oxygen Ozone Therapy in the Treatment of Chronic Obstructive Pulmonary Disease: An Integrative Approach. Am J Clin Exp Med. 2014;2(2):9-13. DOI:10.11648/j.ajcem.20140202.11
- [Background] Vinnik IS, Salmina AB, Tepliakova OV, Drobushevskaia AI, Pozhilenkova EA, Morgun AV, Shapran MV, Kovalenko AO. [The results of combined ozone therapy using in complex treatment of soft tissues infections in patients with diabetes mellitus type II]. Khirurgiia (Mosk). 2015;(2):63-69. doi: 10.17116/hirurgia2015263-69. Russian. PMID 26031822
- [Background] Delgado-Roche L, Riera-Romo M, Mesta F, Hernandez-Matos Y, Barrios JM, Martinez-Sanchez G, Al-Dalaien SM. Medical ozone promotes Nrf2 phosphorylation reducing oxidative stress and pro-inflammatory cytokines in multiple sclerosis patients. Eur J Pharmacol. 2017 Sep 15;811:148-154. doi: 10.1016/j.ejphar.2017.06.017. Epub 2017 Jun 13. PMID 28623000
- [Background] Niu T, Lv C, Yi G, Tang H, Gong C, Niu S. Therapeutic Effect of Medical Ozone on Lumbar Disc Herniation. Med Sci Monit. 2018 Apr 3;24:1962-1969. doi: 10.12659/msm.903243. PMID 29611536
- [Background] Bocci V. Ozonization of blood for the therapy of viral diseases and immunodeficiencies. A hypothesis. Med Hypotheses. 1992 Sep;39(1):30-4. doi: 10.1016/0306-9877(92)90136-z. PMID 1435389
- [Background] Bocci V. Does ozone therapy normalize the cellular redox balance? Implications for therapy of human immunodeficiency virus infection and several other diseases. Med Hypotheses. 1996 Feb;46(2):150-4. doi: 10.1016/s0306-9877(96)90016-x. PMID 8692040
- [Background] Bassi P, Sbrascini S, Mattassi R, D'Angelo F, Franchina A. [Ozone in the treatment of herpes zoster]. Riv Neurobiol. 1982 Jul-Dec;28(3-4):328-33. No abstract available. Italian. PMID 7187109
- [Background] Gierek-Lapinska A, Antoszewski Z, Myga B, Skowron J. [Preliminary report on using therapeutic ozone in infectious conjunctivitis and keratitis and in corneal degeneration]. Klin Oczna. 1992 May-Jun;94(5-6):137-8. Polish. PMID 1453672
- [Background] Mandzhgaladze NR, Kharebava ER, Didia TsG, Ardzhevanishvili MD, Gudzhabidze MV, Chigiashvili TsN. [Influence of intravenous ozone treatment on the level of different specificity antibodies]. Georgian Med News. 2006 Sep;(138):93-5. Russian. PMID 17057311
- [Background] Huang J, Huang J, Xiang Y, Gao L, Pan Y, Lu J. [Topical ozone therapy: An innovative solution to patients with herpes zoster]. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2018 Feb 28;43(2):168-172. doi: 10.11817/j.issn.1672-7347.2018.02.011. Chinese. PMID 29559601
- [Background] Jiao XJ, Peng X. [Clinilal study of medical ozone therapy in chronic hepatitis B of 20 patients]. Zhonghua Shi Yan He Lin Chuang Bing Du Xue Za Zhi. 2008 Dec;22(6):484-5. Chinese. PMID 19544653
- [Background] Chernyshev AL, Filimonov RM, Karasev AV, Neronov VA, Maksimov VA. [Combined treatment including ozonotherapy of patients with viral hepatitis ]. Vopr Kurortol Fizioter Lech Fiz Kult. 2008 May-Jun;(3):19-22. Russian. PMID 18655281
- [Background] Neronov VA. [Experience with the use of ozone for the treatment of chronic viral hepatitis]. Vopr Kurortol Fizioter Lech Fiz Kult. 2009 Nov-Dec;(6):14-7. Russian. PMID 20017375
- [Background] Cespedes-Suarez J, Martin-Serrano Y, Carballosa-Peña MR, Dager-Carballosa DR . Response of patients with chronic Hepatitis B in one year of treatment with Major Autohemotherapy. J Ozone Ther. 2018:2(3) DOI:10.7203/jo3t.2.3.2018.11459
- [Background] Zaky S, Kamel SE, Hassan MS, Sallam NA, Shahata MA, Helal SR, Mahmoud H. Preliminary results of ozone therapy as a possible treatment for patients with chronic hepatitis C. J Altern Complement Med. 2011 Mar;17(3):259-63. doi: 10.1089/acm.2010.0016. PMID 21417811
- [Background] Mawsouf MN, Tanbouli TT, Viebahn-Hänsler R. Ozone therapy in patients with viral Hepatitis C: Ten Years' Experience. Ozone Sci Eng. 2012;34(6):451-458. DOI:10.1080/01919512.2012.720161
- [Background] Ibrahim AM, Elkot RA, Khashaba SA. Successful Treatment of Multiple Common Warts With Intralesional Ozone. Dermatol Surg. 2020 Jul;46(7):928-933. doi: 10.1097/DSS.0000000000002174. PMID 31584525
- [Background] Cespedes-Suarez J, Martin-Serrano Y, Carballosa-Peña MR, Dager-Carballosa DR. The immune response behavior in HIV-AIDS patients treated with Ozone therapy for two years. J Ozone Ther. 2019:2(3). DOI:10.7203/jo3t.2.3.2018.11458